CLINICAL TRIAL: NCT05292872
Title: Replicate Studies Evaluating the Effectiveness of Obeticholic Acid on Hepatic Real-World Outcomes in Patients With Primary Biliary Cholangitis
Brief Title: Real-World Data Study to Evaluate the Effectiveness of OCA on Hepatic Outcomes in PBC Patients
Acronym: HEROES PBC
Status: Completed | Type: Observational
Sponsor: Intercept Pharmaceuticals (Industry)
Collaborators: Target RWE (Industry); Syneos Health (Other); Komodo Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 747-405
Record Dates: First submitted 2022-03-04; First posted 2022-03-23 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary Biliary Cholangitis; Primary Biliary Cirrhosis; PBC; Hepatic Impairment; Liver
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OCA-treated: PBC participants with a history of UDCA failure (inadequate response, intolerance, or discontinuation) who initiated Obeticholic acid (OCA) in the study window.
- Non-OCA Treated: PBC participants with a history of UDCA failure who were eligible but not treated with OCA (or off-label fibrates) in the study window.

SUMMARY:
This is an observational, retrospective cohort study of patients with primary biliary cholangitis (PBC) who failed ursodeoxycholic acid (UDCA) treatment, using a real-world data source, the Komodo Health United States (US) claims database. The study is designed to evaluate the effectiveness of obeticholic acid (OCA). All patients who meet diagnostic criteria for PBC in the database between 01 Jun 2015 and 31 Dec 2021 and who meet all eligibility criteria were considered for this study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Definite or probable PBC diagnosis
2. Inadequate response or intolerance to UDCA
3. Age ≥18 years at the index date
4. Continuous enrollment and evaluable data for at least 12 months before the index date (inclusive)

Key Exclusion Criteria:

1. History or presence of other concomitant liver diseases
2. History of non-skin malignancy or melanoma
3. History of HIV
4. Medical conditions that may cause non-hepatic increases in ALP
5. Patients with laboratory values indicative of hepatic decompensation or significant hepatobiliary injury
6. History of liver transplant
7. Evidence of fenofibrate, or bezafibrate use
8. History or presence of hepatic decompensating events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet diagnostic criteria in each database between 01 Jun 2015 and 31 Dec 2021 and who meet the eligibility criteria were considered for these studies.
Sampling Method: Non-Probability Sample
Enrollment: 4577 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Szczech, MD, Study Director — Intercept Pharmaceuticals
Locations (1):
- Intercept Pharmaceuticals, Inc, San Diego, California, United States

REFERENCES:
- [Derived] Brookhart MA, Mayne TJ, Coombs C, Breskin A, Ness E, Bessonova L, Chu YJ, Li J, Fried MW, Hansen BE, Kowdley KV, Jones D, Mells G, Trivedi PJ, Hiu S, Kareithi DN, Wason J, Smith R, Seeger JD, Hirschfield GM. Hepatic real-world outcomes with obeticholic acid in primary biliary cholangitis (HEROES): A trial emulation study design. Hepatology. 2025 Jun 1;81(6):1647-1659. doi: 10.1097/HEP.0000000000001174. Epub 2025 Jan 3. PMID 39630028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the United States (US) and data was analyzed from Komodo Health claims database between 01 Jun 2015 to 31 Dec 2021.
Pre-assignment Details: Participants were included if, between 01Jun2015 and 31Dec2021, they met criteria for PBC diagnosis: At least 1 inpatient claim with an associated PBC International Classification of Diseases (ICD)-10 code, or at least 2 outpatient claims separated by >1 day with a PBC ICD-9 or ICD-10 code. Patient records (indexes) were selected from a healthcare database. The unit of analysis were indexes, not participants. Analysis was conducted using weighted index methods.
Units Other Than Participants: Indexes
Groups:
- OCA-treated: PBC participants with a history of Ursodeoxycholic acid (UDCA) failure (inadequate response, intolerance, or discontinuation) who initiated Obeticholic acid (OCA) in the study window were included.
- Non-OCA Treated: PBC participants with a history of UDCA failure who were eligible but not treated with OCA for the study. This was a real-world study, and it was conducted in a population of participants selected from a database using weighted index methods.
Period: Overall Study
Arm/Group | OCA-treated | Non-OCA Treated
Started (The unit of analysis is Indexes. The non-OCA group shows the weighted number of units.) | 403; 403 Indexes | 4174; 405 Indexes
Completed | 403; 403 Indexes | 4174; 405 Indexes
Not Completed | 0; 0 Indexes | 0; 0 Indexes

BASELINE CHARACTERISTICS:
Population: Weighted index population. The SMR weights were used to create a pseudo-population of non-OCA-treated indexes with the same covariate distribution as the OCA-treated participants at the time of OCA initiation and weighted standardized mean differences (SMDs) were computed. This was a real-world study, and it was conducted in a population of patients selected from a databased using weighted index methods" The unit of analysis is Indexes.
Units Other Than Participants: Indexes
Groups:
- OCA-treated: PBC participants with a history of UDCA failure (inadequate response, intolerance, or discontinuation) who initiated OCA in the study window were included.
- Total: Total of all reporting groups
Arm/Group | OCA-treated | Non-OCA Treated | Total
Number analyzed (Participants) | 403 | 4174 | 4577
Number analyzed (Indexes) | 403 | 405 | 808
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.213 (10.580) | 55.859 (12.599) | 56.036 (11.638)
Sex: Female, Male [Count of Units; unit: Indexes]
  Female | 369 | 369 | 738
  Male | 34 | 36 | 70
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region [Count of Units; unit: Indexes]
  Northeast | 82 | 84 | 166
  Midwest | 38 | 38 | 76
  West | 97 | 106 | 203
  South | 186 | 175 | 361
  Territory | 0 | 1 | 1
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Risk of the First Event of the Composite Events
Description: The primary analysis outcome was assessed with hazard ratio (HR) comparing hazard of first event of the composite endpoint among OCA-treated participants and SMR-weighted non-OCA-treated PBC participants indexes. It included all-cause death, liver transplant, hospitalization for hepatic decompensation based on first occurrence of: variceal bleed, ascites (including hepatic hydrothorax and spontaneous bacterial peritonitis) and hepatic encephalopathy. OCA-treated indexes were censored 90 days after OCA discontinuation, or if fibrates were initiated. Control indexes were censored if a participant-initiated OCA therapy, initiated fibrate therapy, reinitiated UDCA for participants who had discontinued UDCA for >6 months, or end of study period (31 Dec 2021), whichever came first. The 2.5th and 97.5th percentile of nonparametric bootstrap samples were used to estimate 95% CI for HR and to perform a test of hypothesis. Risk is presented using the number of composite event and components.
Time Frame: Up to 67 months
Population: Weighted index population. The unit of analysis is Indexes.
Measure: Number; unit: Events during the study period
Units Other Than Participants: Indexes
Arm/Group | OCA-treated | Non-OCA Treated
Number analyzed (Participants) | 403 | 4174
Number analyzed (Indexes) | 403 | 405
Events during the study period | 8 | 32
Statistical Analysis 1: Comparison: OCA-treated vs Non-OCA Treated; Test type: Superiority; p < .001, Nonparametric bootstrap approach — 1-sided p-values are proportion of bootstrap replicates exceeding null (defined as a HR of 1) in each direction), and the two-tailed p-value is twice the smaller of one-tailed p-values. A two-tailed p-value was calculated for HR using this method; Hazard Ratio (HR) = 0.370, 95% CI 2-sided [0.143 to 0.752]

2. Secondary Outcome: Risk of Death
Description: The primary source for death was the Social Security Death Index (SSDI) along with obituary search, which was compared to Komodo Health claims and LabCorp/Quest laboratory data. The secondary objectives were to estimate the effect of OCA treatment versus non-OCA treatment on each component of the composite endpoint, with the same censoring rule applied as in the primary composite endpoint. Risk is presented using the the number of all-cause death within the risk period (prior to censoring).
Time Frame: Up to 67 months
Population: Weighted index population. The unit of analysis is Indexes.
Measure: Number; unit: Events during the study period
Units Other Than Participants: Indexes
Arm/Group | OCA-treated | Non-OCA Treated
Number analyzed (Participants) | 403 | 4174
Number analyzed (Indexes) | 403 | 405
Events during the study period | 2 | 9

3. Secondary Outcome: Risk of Liver Transplantation
Description: The primary source for liver transplant was the Organ Transplant Network (OPTN) transplant registry. Risk is presented using the number of liver transplantation.
Time Frame: Up to 67 months
Population: Weighted index population. The unit of analysis is Indexes.
Measure: Number; unit: Events during the study period
Units Other Than Participants: Indexes
Arm/Group | OCA-treated | Non-OCA Treated
Number analyzed (Participants) | 403 | 4174
Number analyzed (Indexes) | 403 | 405
Events during the study period | 2 | 12

4. Secondary Outcome: Risk of Hospitalization for Hepatic Decompensation
Description: The primary source for hospitalization for hepatic decompensation were Komodo Health claims. Risk is presented using the number of hospitalization for hepatic decompensation.
Time Frame: Up to 67 months
Population: Weighted index population. The unit of analysis is Indexes.
Measure: Number; unit: Events during the study period
Units Other Than Participants: Indexes
Groups:
- OCA-treated: PBC participants with a history of UDCA failure (inadequate response, intolerance, or discontinuation) who initiated OCA in the study window (01-Jun-2015 and 31-Dec-2021) were included.
Arm/Group | OCA-treated | Non-OCA Treated
Number analyzed (Participants) | 403 | 4174
Number analyzed (Indexes) | 403 | 405
Events during the study period | 6 | 23

ADVERSE EVENTS:
Time Frame: Up to 67 months
Description: This is an observational real-world data study to evaluate the effectiveness of OCA on hepatic outcomes in participants with PBC and the study did not plan to evaluate safety endpoints. The unit of analysis is Indexes. For all-cause mortality, numbers of all death cases during the whole study period (no censoring applied) are presented.
Arm/Group | OCA-treated | Non-OCA Treated
All-Cause Mortality (participants affected / at risk) | 12/403 | 17/405
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This is an observational real-world data study to evaluate the effectiveness of OCA on hepatic outcomes in participants with PBC and the study did not plan to evaluate safety endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT05292872/Prot_SAP_000.pdf